CLINICAL TRIAL: NCT01972464
Title: Progesterone for Postpartum Smokers: Feasibility, Breastfeeding and Infant Safety
Brief Title: Progesterone for Smoking Relapse Prevention Following Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1305012130; R21DA035924 (NIH)
Record Dates: First submitted 2013-10-17; First posted 2013-10-30 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Tobacco Use Disorder
Keywords: Progesterone; Placebo; Postpartum; Tobacco; Pregnancy
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): In this group women will receive a placebo pill which will appear similar to progesterone and will be inert.
  Interventions: Drug: Placebo
- Progesterone (Experimental): In this group women will receive oral micronized progesterone twice a day.
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — oral micronized progesterone
  Arms: Progesterone
Drug: Placebo
  Arms: placebo

SUMMARY:
Smoking is the main preventable cause of mortality in Western countries, contributing to over 430,000 deaths a year in the U.S. alone. Clinical and epidemiological studies show that women often decrease smoking in pregnancy, when progesterone levels are high. However, at least half resume pre-pregnancy smoking levels within weeks after delivery and when progesterone levels drop.

Data from preclinical and clinical studies suggest that progesterone may be effective in preventing relapse to smoking in non-postpartum women. Prior work has shown that progesterone decreases both craving for cigarettes and the subjective rewarding effects of smoking among recently abstinent female smokers. These findings led us to hypothesize that progesterone may have efficacy as a relapse prevention treatment for postpartum women.

We propose an 8-week, randomized pilot study to evaluate the safety and initial efficacy of progesterone. This will be a feasibility study that will compare progesterone to placebo for relapse prevention in 40 postpartum smokers. We will assess the feasibility and safety, including the potential effects on breastfeeding and infants exposed via breast milk, in addition to 7-day point prevalence of smoking abstinence after 8 weeks of treatment and at follow-up, 3-months after the end of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Need to be within 3 weeks of delivery because relapse to smoking happens early after childbirth
* Aged 18 to 42 years
* history of smoking, with smoking and other nicotine product abstinence achieved in the final two months of pregnancy and at delivery
* In good health as verified by medical history
* Using acceptable birth control methods other than hormonal contraceptives that contain progestins
* Have biologically confirmed abstinence from tobacco and other nicotine products at randomization

Exclusion Criteria:

* A history of major medical illnesses including liver diseases, suspected or known malignancy, thrombophlebitis, liver failure, or other medical conditions that the physician investigator deems will make study participation unsafe for the subject
* Current or past history bipolar disorder or schizophrenia or current diagnosis of major depression, panic disorder or post-traumatic stress disorder
* Dependence on and/or abuse of alcohol or other drugs of abuse in the month prior to randomization into the trial
* the presence of suicidal or homicidal ideation, or significant impairment of social or occupational functioning, either at study baseline during the evaluation process, or during participation in the trial
* inability to speak Spanish or English (our group is bilingual)
* plans to move out of the area within 8 months after study screening since this will make follow-up difficult
* Inability to understand study procedures or provide informed consent
* Currently undergoing treatment with another pharmacological agent for smoking cessation
* pending legal case that may result in incarceration since this would force abstinence and impede follow-up;
* Pending case with child protective services that might lead removal of infant from mother's custody, as this would impede breastfeeding and infant follow-up
* Unwilling to accept randomization
* Subsequent pregnancy since that would be another source of progesterone
* An acute general medical condition that would require imminent re-hospitalization since this would enforce abstinence (women may be randomized if they are discharged and still within the recruitment window)
* Allergy to progesterone or peanuts (vehicle for micronized progesterone)
* Currently undergoing treatment with ketoconazole or any other known strong CYP3A4 inhibitors

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Forray, MD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine Dpt of Psychiatry, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began January 2014 and final data collection occurred August 2016. We accepted study referrals and conducted on-site clinic screening assessments in three academic obstetrics clinics associated with Yale New Haven Hospital.
Pre-assignment Details: We screened 90 pregnant women who were current smokers intending to quit prior to 32 weeks gestation; 26 were ineligible because they were still smoking at 32 weeks gestation (n=12) or did not meet other eligibility criteria (n=14); 23 were eligible but not randomized because they declined to participate (n=8) or were out of contact (n=15).
Groups:
- Placebo: In this group women will receive a placebo pill which will appear similar to progesterone and will be inert.
  Placebo
- Progesterone: In this group women will receive oral micronized progesterone twice a day.
  Progesterone
Period: Treatment Period (Week 1 Through Week 8)
Arm/Group | Placebo | Progesterone
Started | 19 | 22
Completed | 16 | 18
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 3
Not completed — Patient Relocated | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: 3-Month Follow-Up (Week 20)
Arm/Group | Placebo | Progesterone
Started | 16 | 18
Completed | 15 | 17
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Progesterone | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.3) | 26.2 (4.9) | 25.8 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black, non-Latina | 13 | 9 | 22
  Race/Ethnicity: Latina | 4 | 11 | 15
  Race/Ethnicity: White, non-Latina | 1 | 2 | 3
  Race/Ethnicity: More than one race, non-Latina | 1 | 0 | 1
Education level [Count of Participants; unit: Participants]
  <High school degree | 3 | 6 | 9
  High school degree | 9 | 13 | 22
  Some college (no degree) | 7 | 3 | 10
Lives with spouse or partner [Count of Participants; unit: Participants]
  Yes | 10 | 10 | 20
  No | 9 | 12 | 21
Lives with smoker [Count of Participants; unit: Participants] — Population: 4 participants did not report this information
  Participants
    number analyzed (Participants) | 16 | 21 | 37
    Yes | 8 | 10 | 18
    No | 8 | 11 | 19
Parity [Count of Participants; unit: Participants]
  1 | 3 | 8 | 11
  2 | 8 | 4 | 12
  3 | 4 | 7 | 11
  4+ | 4 | 3 | 7
Pre-quit number of cigarettes per day [Mean (Standard Deviation); unit: participants] — Population: 6 participants did not report this information
  participants
    number analyzed (Participants) | 16 | 19 | 35
    (all) | 7.1 (3.3) | 6.2 (4.3) | 6.6 (3.9)
Pre-quit smoking level [Count of Participants; unit: Participants]
  ≤10 cigarettes/day | 17 | 17 | 34
  10 cigarettes/day | 2 | 5 | 7
Breastfeeding intentions [Count of Participants; unit: Participants]
  Breastfeed exclusively | 4 | 9 | 13
  Breasefeed and formula feed | 10 | 11 | 21
  Formula feed exclusively | 4 | 2 | 6
  Unsure | 1 | 0 | 1
Feeding method at week 2 visit [Count of Participants; unit: Participants]
  Breastfeed exclusively | 0 | 6 | 6
  Breasefeed and formula feed | 3 | 5 | 8
  Formula feed exclusively | 14 | 7 | 21
  Missing | 2 | 4 | 6
Fagerstrom Test for Nicotine Dependence [Count of Participants; unit: Participants]
  Low dependence | 6 | 7 | 13
  Low to moderate dependence | 9 | 11 | 20
  Moderate dependence | 4 | 4 | 8
  High dependence | 0 | 0 | 0
Questionnaire on Smoking Urges (QSU)-Brief Score [Mean (Standard Deviation); unit: units on a scale] — Scale is scored from 10 to 70. Higher scores indicate more severe symptoms.
  units on a scale | 15.6 (15.4) | 18.0 (12.2) | 16.9 (13.7)
Edinburgh Postnatal Depression Scale Score [Mean (Standard Deviation); unit: units on a scale] — Scale is scored from 0 to 30. Higher scores indicate more severe symptoms.
  units on a scale | 3.8 (4.9) | 3.0 (4.5) | 3.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Progesterone as a Relapse Prevention Intervention for Postpartum Women With Pre-conception Smoking: Adherence to Treatment
Description: Feasibility will be shown by high adherence to treatment condition assessed by doses of study medication taken
Time Frame: 8 weeks
Population: Adherence to treatment as measured by mean (SD) doses of study medication taken by women in each arm of the study.
Measure: Mean (Standard Deviation); unit: doses of medication
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 19 | 22
doses of medication | 84.5 (38.3) | 76.0 (42.0)

2. Primary Outcome: Feasibility of Progesterone as a Relapse Prevention Intervention for Postpartum Women With Pre-conception Smoking: Retention
Description: Feasibility in retention will be shown by at least 70% of women randomized to the progesterone group reamaining in the study at the 3-month follow-up
Time Frame: From randomization to 3-month follow-up: up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 19 | 22
Participants | 15 | 17

3. Secondary Outcome: 7-day Point Prevalence of Abstinence at End of Treatment (Week 8)
Description: Abstinence was defined as self-report of no smoking in the past 7 days confirmed by a negative urine cotinine test (urine cotinine <100 ng/ml).
Time Frame: Week 8 of the trial period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 19 | 22
Participants | 6 | 10
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Null hypothesis- odds of week 8 point prevalence abstinence were equal between placebo and progesterone group; Test type: Superiority; p = 0.39, Regression, Logistic — a priori threshold for statistical significance = 0.05; adjusted for age (18-25 years versus >25 years) and pre-quit smoking level (<10 versus >10 cigarettes per day); Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.48 to 6.52] — OR represents of odds of abstinence in progesterone group versus placebo group

4. Post Hoc Outcome: Time to Relapse
Description: The Outcome Measure is reporting the time in weeks to relapse
Time Frame: baseline through 3-month post trial follow-up
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 19 | 22
weeks | 4 [2 to 10] | 10 [3 to NA] — For the Inter-Quartile Range in the progesterone group, > than 25% of the data were right censored so 75th percentile could not be calculated
Statistical Analysis 1: Comparison: Placebo vs Progesterone; Test type: Superiority; p = 0.41, Regression, Cox — a priori threshold = 0.05; Adjusted for age and pre-quit smoking level; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.66 to 3.38] — Hazard ratio is placebo / progesterone

5. Post Hoc Outcome: Questionnaire on Smoking Urges (QSU)-Brief Score
Description: Scale is scored from 10 to 70. Higher scores indicate more severe symptoms
Time Frame: treatment period; baseline through week 8, measured weekly
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Progesterone
Number analyzed (Participants) | 19 | 22
units on a scale
  baseline | 15.6 (15.4) | 18.0 (12.2)
  week 1 | 13.3 (5.6) | 14.5 (10.5)
  weeek 2 | 14.1 (7.8) | 13.7 (7.5)
  week 3 | 15.5 (9.7) | 14.5 (9.1)
  week 4 | 18.3 (10.6) | 12.2 (3.8)
  week 5 | 15.7 (6.8) | 13.8 (8.5)
  week 6 | 17.9 (10.0) | 12.1 (5.1)
  week 7 | 17.2 (8.6) | 10.6 (2.4)
  week 8 | 21.4 (17.5) | 10.4 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Progesterone; null hypothesis rate of change in QSU-brief scores were equal between treatment groups; Test type: Superiority; p < 0.001, general estimating equation; adjusted for age & pre-quit smoking level; specified a gamma distribution, log link, autoregressive correlation structure; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.86 to 0.96] — risk ratio is progesterone versus placebo

ADVERSE EVENTS:
Time Frame: baseline through teh 8 week trial period and the 3-month follow-up visit
Arm/Group | Placebo | Progesterone
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 3/19 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Progesterone (N=22)
headache (General disorders) | 1 (1) | 0 (0) — headache
feeling Warm (General disorders) | 1 (2) | 0 (0) — feeling warm
Itching (General disorders) | 1 (1) | 0 (0) — Itching
abnormal pap smear (Reproductive system and breast disorders) | 0 (0) | 1 (1) — abnormal pap smear; repeat pap smear was negative
heavy menses (Reproductive system and breast disorders) | 0 (0) | 1 (1) — heavy menses during first cycle following delivery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No